CLINICAL TRIAL: NCT01812590
Title: Acute Exercise and Pancreatic Endocrine Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Solomon, Senior Researcher, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Ex-Panc
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise

ARMS (2):
- Resting Trial (No Intervention): Pancreatic endocrine function will be determined the morning following a day where no exercise is performed
- Exercise Trial (Experimental): Pancreatic endocrine function will be determined the morning following a day where a 1-hour aerobic exercise is performed at 65% of pre-determined HRmax (maximal heart rate measured during an incremental work-load exercise test to volitional exhaustion)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise
  Arms: Exercise Trial

SUMMARY:
Subjects with type 2 diabetes will be stratified into two-quantiles based on ambient hyperglycemia (fasting glucose and HbA1c) and then the effects of a single aerobic exercise bout (1-hour at 50%VO2max) on pancreatic endocrine function will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis with type 2 diabetes, or newly detected in our screening procedures
* Age 30-70 years
* BMI 20-40 kg/m2

Exclusion Criteria:

* Treatment with insulin
* Contraindication to exercise as determined by ECG
* Pregnancy
* Active weight loss in the previous 6 months
* Actively engaged in exercise training programs
* Evidence of chronic pulmonary, cardiovascular, hepatic, renal, or hematological disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Pancreatic endocrine function | 24-hours following a period of rest/exercise
  Insulin and glucagon secretory responses to intravenous glucose (hyperglycemic clamp 5.4 mmol/l above basal), glucagon-like peptide-1 (0.5 pmol/kg/min), and arginine (5 g injection) will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark